CLINICAL TRIAL: NCT04111289
Title: Effect of Upstream High Bolus Dose of Tirofiban in Primary PCI for the Patients With STEMI on Short Term Outcome
Acronym: TISP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Qaood Mohammed, Principel investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tirofiban in STEMI patient
Record Dates: First submitted 2019-09-29; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: High Bolus Dose of Tirofiban

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient received upstream high bolus dose of tirofiban (Active Comparator): * After consenting for primary PCI ,the patient will be assigned to one arm ( either upstream high bolus dose IV before going to cath lab or selective downstream administration according to operator discretion )
  * Administration of tirofiban (25 ug/kg bolus and 0.15 ug/kg/min maintenance infusion)
  * Randomization will be performed by Microsoft Excel where random order will be generated for the study population
  Interventions: Drug: -Administration of tirofiban (25 ug/kg bolus and 0.15 ug/kg/min maintenance infusion)
- Patients did not receive upstream high bolus dose of tirofiban (Active Comparator): Patient receive tirofiban downstream selectively according to operator discretion
  Interventions: Drug: -Administration of tirofiban (25 ug/kg bolus and 0.15 ug/kg/min maintenance infusion)

INTERVENTIONS:
Drug: -Administration of tirofiban (25 ug/kg bolus and 0.15 ug/kg/min maintenance infusion) — * After consenting for primary PCI ,the patient will be assigned to one arm ( either upstream high bolus dose IV before going to cath lab or selective downstream administration according to operator discretion )
  * Administration of tirofiban (25 ug/kg bolus and 0.15 ug/kg/min maintenance infusion)
  * Randomization will be performed by Microsoft Excel where random order will be generated for the study population

SUMMARY:
The goal of the study to investigate the impact of upstream HBD of Tirofiban on short outcome of STEMI patient.

DETAILED DESCRIPTION:
* Primary percutaneous coronary intervention (PPCI) is the gold standard of treatment of ST segment elevation myocardial infarction (STEMI).1 PPCI restores thrombolysis in myocardial infarction flow 3 (TIMI 3) in over 90% of patients. However ,there remains a small proportion of patients, who continue to exhibit overt impairment of myocardial reperfusion despite successful opening of infarct related epicardiual artery (IRA). This phenomenon is called no-reflow, which is largely because of severe microvascular obstruction (MVO).
* Belonging to the class of glycoprotein IIb/IIIa inhibitors (GPIs), tirofiban, can be useful in primary PCI for acute coronary syndrome (ACS).1,2The administration of tirofiban is an efficacious treatment option to reduce ischemic events in patients with The ACS and/or those undergoing PCI.2,3 In most guidelines, abciximab is recommended as the drug of first choice4 due to the finding that tirofiban is less effective than abciximab in platelet inhibition within 60 min of intravenous administration. However, some recent systemic reviews of randomized trials have not demonstrated obvious difference between smGPIs (eptifibatide or tirofiban) and abciximab in terms of angiographic, electrocardiographic, and clinical outcomes of patients undergoing primary PCI.5,6 Tirofiban may provide similar efficacy with an improved safety profile when compared with abciximab, particularly with a high-dose bolus regimen.7,8 In the new guideline, the recommended class of smGPIs has changed from IIb to IIa, but tirofiban remains with a pre-PCI indication of IIb, B.4 Although early treatment was associated with a significantly better TIMI flow and superior TIMI myocardial perfusion grades (TMPG) in some trials,9,10 no difference in clinical outcome was found between the 2 strategies in later study.11 One potential cost of administration of GPIs could be increased bleeding, although both major bleeding and minor bleeding rate are low in the tirofiban-treated patients..

ELIGIBILITY:
Inclusion Criteria:

* - Acute STEMI patient within 12 hours of chest pain

Exclusion Criteria:

* -previous infarction in the same infarct- related artery
* ISR
* Resistent cardiogenic shock
* Known CKD with Cr cl less than 60 ml/min
* Uncontrolled HTN more than 180/110 mmHg
* Suspected aortic dissection
* Traumatic or prolonged CPR
* Severe trauma or major surgery within 3 month
* Active peptic ulcer within past 3 month
* Known history of coagulopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-01-28 (Estimated)

PRIMARY OUTCOMES:
Primary (main): | 40 days
  Angiographic result (TIMI flow & MB) after PPCI.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Qaood, Principal Investigator — Assiut University